CLINICAL TRIAL: NCT07056634
Title: The Effects of Nature-Based Activity vs. Indoor Exercise on Cognitive, Psychological, and Physiological Health: A Randomized Controlled Trial
Brief Title: The Effects of Nature-Based Activity vs. Indoor Exercise on Cognition, Psychological, and Physiological Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Ministry of Higher Education, Malaysia (Other)
Responsible Party: Principal Investigator, Tan Kok Wei, Dr., University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UoRM REC 2025/05; FRGS/1/2023/SS09/READING/03/1 (Other Grant/Funding Number: University of Reading Malaysia)
Record Dates: First submitted 2025-06-19; First posted 2025-07-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-06

CONDITIONS: Psychological Well Being; Cognitive Performance
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Nature Engagement (Experimental): Outdoor walking in a designated urban park, 3 times/week for 4 weeks, 30 minutes/session
  Interventions: Behavioral: Active Nature Engagement
- Passive Nature Engagement (Experimental): Sitting quietly and observing nature, with grounding exercise, 3 times/week for 4 weeks, 30 minutes/session
  Interventions: Behavioral: Passive Nature Engagement
- Indoor Exercise (Active Comparator): Treadmill walking indoors under controlled conditions, 3 times/week for 4 weeks, 30 minutes/session
  Interventions: Behavioral: Indoor Exercise
- Control (No Intervention): No exposure to intervention between baseline and post-test

INTERVENTIONS:
Behavioral: Active Nature Engagement — Participants in this group will walk at a comfortable pace for 30 minutes in an urban park, three times per week for four weeks. They will be guided to focus on their surroundings using a grounding exercise (e.g., noticing sights, sounds, and smells) and instructed not to use mobile phones or listen to music during the walk.
  Arms: Active Nature Engagement
Behavioral: Passive Nature Engagement — Participants in this group will sit quietly for 30 minutes in a designated spot within an urban park, three times per week for four weeks. They will engage in grounding exercises and draw aspects of the natural environment. Participants will be instructed not to use mobile phones or listen to music during the walk.
  Arms: Passive Nature Engagement
Behavioral: Indoor Exercise — Participants will be asked to walk on a treadmill in an indoor room without windows for 30 minutes. The treadmill will be set to the speed that match the average pace in nature walk group (approximately 3 km/hr). The speed could be adjusted by the participant if needed, but kept within the range of 2.6 km/hr to 4.6 km/hr. Participants will be asked to not use their phones or listen to music.
  Arms: Indoor Exercise

SUMMARY:
This randomized controlled trial aims to investigate the comparative effects of nature-based versus indoor exercise interventions on cognitive performance, psychological well-being, and physiological stress in Malaysian adults. Participants will be randomly assigned to one of four groups: (1) active nature engagement (walking outdoors), (2) passive nature engagement (seated outdoor observation), (3) indoor treadmill walking, or (4) a no-intervention control group. The study will examine changes in attention, working memory, affect, blood pressure, body composition, and salivary cortisol across baseline, mid-point, and post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing
* Physically fit - able to walk unassisted for at least 30 minutes

Exclusion Criteria:

* Participants with limited mobility that prevents outdoor activities
* Participants who do not have adequate comprehension in English necessary to participate in measurement of outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained attention | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Sustained attention to response task (SART) will be used to measure sustained attention. Participants will be presented with a series of single digits (1-9) displayed one at a time on a computer screen. The digit appears in a random order at a fixed interval. They will be instructed to press the spacebar as quickly as possible every time they see any digit except the target digit (i.e., the digit 3). Participants are instructed to withhold their response when the target digit appears.
Salivary cortisol | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Participants' salivary cortisol will be collected using the passive drool method in sampling tubes. The samples were then be sent to the laboratory for measurement of cortisol in saliva, as an indicator for participants' stress level.
Working memory | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Digit span backward (DSB) will be used to measure working memory. A series of digits will be presented sequentially, and the participants will be asked to repeat them in backward order. Sequences were 2 to 8 digits, and there will be a total of 14 trials (with 2 trials for each length).

SECONDARY OUTCOMES:
Executive functioning | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Heart and Flower Task will be used to measure executive functions. The test is comprised of three phases: (1) the congruent trials phase, where participants will be instructed to press the response button corresponding to the side where the heart appeared; (2) the incongruent trial phase, where the participants will be asked to press the opposite response button corresponding to the side where the flower appeared and; (3) the mixed phase, comprising a mix of congruent and incongruent trials. During all phases, stimuli were displayed for 750ms, and participants will have 1 second to respond accurately while holding instructions in mind, which requires a working memory function. Additionally, cognitive flexibility will be necessary during phase three, where participants will have to switch rules flexibly and inhibit responding on the same side when the flower appeared in phases two and three.
Creativity | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Alternate Uses Task (AUT) will be used to evaluate divergent creative thinking and cognitive flexibility. Participants will be provided with two items (i.e., a tennis ball, a coffee cup)) and they will be required to come up with as many alternative uses for it as they can, in 2 minutes. The responses will be evaluated on four components: (1) fluency, refers to the total number of non-repeated, appropriate responses, and any responses that were infeasible, vague, or similar to the common use will be discarded; (2) flexibility, refers to the number of different topics or categories of responses; (3) elaboration, refers to the level of detail and development of each idea, measured by the average number of words per response; (4) originality, refers to the statistically uncommon response when compared to the overall data set.
Positive and negative affect | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Positive and negative affect schedule (PANAS) is a self-report tool that consists of 20 items, where 10 items measure positive affect (PA) and 10 items measure negative affect (NA). Participants will rate their affect over the past week on a 5-point Likert scale from 1 (not at all) to 5 (extremely). The scores for PA and NA are calculated by adding up the items that measure the respective constructs, with scores ranging from 10 to 50. Higher scores indicate higher levels of PA or NA.
Stress level | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Perceived stress scale (PSS-10) will serve as a subjective measure of participants' stress levels where it measures the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the past week. Participants will report how they felt on a 5-point Likert scale from 0 (never) to 4 (very often). The score is obtained by summing across all items (with reverse items being reversed-score), higher scores indicate higher levels of perceived stress.
Blood pressure | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  The blood pressure (BP) of participants (both diastolic and systolic BP) will be measured using a standard sphygmomanometer. A sphygmomanometer is a non-invasive measurement of bodily arousal.
Body weight | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Weight measured using TANITA body composition scale. Reported in kg.
Muscle mass | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Measured via TANITA body composition scale, and reported in kg.
Body fat percentage | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Estimated body fat proportion measured using TANITA body composition scale, reported in %.
Visceral fat level | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Rating provided by TANITA body composition scale indicating estimated visceral fat level. This will be reported in unitless scale rating from 1-59.
Total body water percentage | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Percentage of body weight that is water, measured by TANITA body composition scale, reported in %.
Daily calorie intake | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Estimated daily caloric requirement provided by TANITA body composition scale based on resting metabolic rate. Reported in kcal/day.
Metabolic age | 1) Baseline (Week 0) 2) Midpoint (Week 2) 3) Post-intervention (Week 4)
  Age estimation based on metabolic profile, as calculated by TANITA body composition scale. Metabolic age will be reported in the unit of 'years'.
Nature relatedness | Baseline (Week 0)
  Nature-relatedness scale (NR-6) will be used to measure one's subjective relatedness to the natural environment. Participants complete 6 items, on a 5-point Likert Scale (with 1 = strongly disagree, 5 = strongly agree). Nature-relatedness will serve as a covariate (will only be measured once).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading Malaysia, Johor Bahru, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: No